CLINICAL TRIAL: NCT04604496
Title: A Phase 1, Non-randomized, Open-label, Single-dose, Parallel Cohort Study to Compare the Pharmacokinetics of PF-06882961 in Adult Participants With Varying Degrees of Hepatic Impairment Relative to Participants Without Hepatic Impairment.
Brief Title: STUDY OF PF-06882961 IN PARTICIPANTS WITH AND WITHOUT VARYING DEGREES OF HEPATIC IMPAIREMENT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: C3421014
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-09

CONDITIONS: Hepatic Impairment; Healthy Volunteers
MeSH Terms: interventions — danuglipron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PF-06882961 participants without Hepatic Impairment (Experimental): This arm includes participants who will receive an oral dose of PF-06882961 20 milligrams (mg) on Day 1
  Interventions: Drug: PF-06882961 20MG
- PF-06882961 participants with mild Hepatic Impairment (Experimental): This arm includes participants who will receive an oral dose of PF-06882961 20 mg on Day 1
  Interventions: Drug: PF-06882961 20MG
- PF-06882961 participants with moderate Hepatic Impairment (Experimental): This arm includes participants who will receive an oral dose of PF-06882961 20 mg on Day 1
  Interventions: Drug: PF-06882961 20MG
- PF-06882961 participants with severe Hepatic Impairment (Experimental): This arm includes participants who will receive an oral dose of PF-06882961 20 mg on Day 1
  Interventions: Drug: PF-06882961 20MG

INTERVENTIONS:
Drug: PF-06882961 20MG — PF-06882961 in 20 mg oral tablet will be administered on Day 1

SUMMARY:
The current study is proposed to evaluate whether there is any clinically meaningful effect of hepatic impairment on the plasma Pharmacokinetic (PK) of PF-06882961

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between the ages of 18 (or the minimum country-specific age of consent if >18) and 70 years, inclusive, at the screening visit:
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Body mass index (BMI) of 17.5 to 38.0 kg/m2, inclusive; and a total body weight >50 kg (110 lb), at the screening visit; with a single repeat assessment of total body weight (and hence BMI), on a separate day permitted to assess eligibility, if needed.

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, prior bariatric surgery, gastrectomy, ileal resection); NOTE: Participants who have undergone cholecystectomy and/or appendectomy are eligible for this study as long as the surgery occurred more than 6 months prior to Screening;
* At screening, participants with a positive result for human immunodeficiency virus (HIV) antibodies, as assessed by sponsor-identified central laboratory, with a single repeat permitted to assess eligibility, if needed;
* A positive COVID-19 test at screening;
* A diagnosis of type 2 diabetes mellitus (T2DM) that is documented by medical history;
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2), or participants with suspected MTC per the investigator's judgement;
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study;
* Use of prior/concomitant therapies
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product used in this study (whichever is longer);
* Participants with known prior participation (ie, randomized and received at least 1 dose of investigational product) in a study involving PF-06882961;
* Participants with ANY of the following abnormalities in clinical laboratory tests at Visit 1, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

HbA1c ≥6.5%; FPG ≥126 mg/Dl; eGFR<60 mL/min/1.73m2;

* A positive urine drug test, for illicit drugs at screening, as assessed by sponsor-identified central laboratory. However, participants in Cohorts 2-4, only, who have been medically prescribed opiates/opioids or benzodiazepines and report the use of these drugs to the investigator at the Screening visit will be allowed to participate; NOTE: repeat urine drug testing is not permitted in this study;
* At screening or Day -1, a positive breath alcohol test, as assessed using kits provided by sponsor-identified central laboratory, with a single repeat on a separate day permitted to assess eligibility, if needed;
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing and until the follow-up contact; 13. History of sensitivity to heparin or heparin-induced thrombocytopenia, only if heparin is used to flush intravenous catheters used during serial blood collections;
* Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol;
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - University of Miami Division of Clinical Pharmacology, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421014

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 29 participants were screened in the study, among whom, 24 participants were treated with PF-06882961 (Danuglipron).
Groups:
- Without Hepatic Impairment: Participants without hepatic impairment received a single, oral dose of PF-06882961 20 mg in the fed state on Day 1.
- Mild Hepatic Impairment: Participants with mild hepatic impairment received a single, oral dose of PF-06882961 20 mg in the fed state on Day 1.
- Moderate Hepatic Impairment: Participants with moderate hepatic impairment received a single, oral dose of PF-06882961 20 mg in the fed state on Day 1.
- Severe Hepatic Impairment: Participants with severe hepatic impairment received a single, oral dose of PF-06882961 20 mg in the fed state on Day 1.
Period: Open Label Treatment
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Follow-Up
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (3.08) | 61.7 (5.85) | 57.7 (7.12) | 56.2 (10.21) | 58.7 (6.89)
Age, Customized [Count of Participants; unit: Participants]
  45-64 Years | 6 | 3 | 5 | 4 | 18
  >=65 Years | 0 | 3 | 1 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 3 | 11
  Male | 3 | 4 | 3 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 3 | 3 | 13
  Not Hispanic or Latino | 2 | 3 | 3 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 5 | 6 | 5 | 22
  Black or African American | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Maximum observed plasma PF-06882961 concentration.
Time Frame: Predose (0 hours), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36 and 48 hours post dose on Day 1.
Population: The analysis population refers to all participants who received at least 1 dose of PF-06882961 and had at least 1 of the pharmacokinetic (PK) parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 23.56 (50) | 31.37 (33) | 51.82 (83) | 78.73 (33)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; Test: the mild hepatic impairment group; Reference: the without hepatic impairment group; Test type: Other — The adjusted ratio and 90% confidence interval from the analysis of variance (ANOVA) model were expressed as percentages; Ratio of adjusted geometric means = 133.17, 90% CI 2-sided [81.97 to 216.37]
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; Test: the moderate hepatic impairment Group; Reference: the without hepatic impairment group; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 219.98, 90% CI 2-sided [135.39 to 357.41]
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; Test: the severe hepatic impairment group; Reference: the without hepatic impairment group; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 334.21, 90% CI 2-sided [205.70 to 543.00]

2. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf)
Description: Area under the plasma PF-06882961 concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: Predose (0 hours), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36 and 48 hours post dose on Day 1.
Population: The analysis population refers to all participants who received at least 1 dose of PF-06882961 and had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL) | 193.4 (83) | 237.3 (34) | 546.7 (116) | 1239 (75)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; Test: the mild hepatic impairment group; Reference: the without hepatic impairment group; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 122.70, 90% CI 2-sided [61.33 to 245.49]
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; Test: the moderate hepatic impairment Group; Reference: the without hepatic impairment group; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 282.73, 90% CI 2-sided [141.32 to 565.66]
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; Test: the severe hepatic impairment group; Reference: the without hepatic impairment group; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 640.78, 90% CI 2-sided [320.27 to 1282.00]

3. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast)
Description: Area under the plasma PF-06882961 concentration-time profile from time 0 extrapolated to the time of the last quantifiable concentration.
Time Frame: Predose (0 hours), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36 and 48 hours post dose on Day 1.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL) | 191.2 (84) | 235.0 (34) | 542.9 (117) | 1217 (73)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; Test: the mild hepatic impairment group; Reference: the without hepatic impairment group; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 122.89, 90% CI 2-sided [61.51 to 245.51]
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; Test: the moderate hepatic impairment Group; Reference: the without hepatic impairment group; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 283.88, 90% CI 2-sided [142.10 to 567.13]
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; Test: the severe hepatic impairment group; Reference: the without hepatic impairment group; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 636.32, 90% CI 2-sided [318.51 to 1271.24]

4. Primary Outcome: Fraction of Unbound Drug in Plasma (fu)
Description: fu = Cu/C (where Cu represents unbound concentration and C represents total concentration).
Time Frame: Predose (0 hours), and 4 hours post dose on Day 1.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
Ratio | 0.02137 (18) | 0.01820 (13) | 0.02059 (21) | 0.02889 (53)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; Test: the mild hepatic impairment group; Reference: the without hepatic impairment group; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 85.19, 90% CI 2-sided [63.60 to 114.10]
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; Test: the moderate hepatic impairment Group; Reference: the without hepatic impairment group; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 96.37, 90% CI 2-sided [71.95 to 129.07]
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; Test: the severe hepatic impairment group; Reference: the without hepatic impairment group; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 135.20, 90% CI 2-sided [100.94 to 181.10]

5. Secondary Outcome: Number of Participants Reporting Treatment-emergent Adverse Events (AEs)
Description: Adverse events (AEs): any untoward medical occurrence in a clinical investigation participant administered a product or medical device, without regard to causality. Treatment-emergent AEs (TEAEs): AEs which occurred for the first time during the effective duration of treatment or AEs that increased in severity during treatment. AEs included SAEs and non-serious AEs. Serious AEs (SAEs) were any untoward medical occurrence at any dose that resulted in death; was life-threatening; required inpatient hospitalization or caused prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions). Treatment-related TEAEs were any untoward medical occurrence attributed to study treatment. Relatedness to study treatment was determined by the investigator.
Time Frame: Baseline to Day 30
Population: All participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  All-causality | 0 | 1 | 2 | 1
  Treatment-related | 0 | 1 | 2 | 1

6. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Protocol-required safety laboratory assessments included: hemoglobin <0.8 x lower limit of normal (LLN), hematocrit <0.8 x LLN, erythrocytes <0.8 x LLN, ery. mean corpuscular volume >1.1 x upper limit of normal (ULN), ery. mean corpuscular hemoglobin >1.1 x ULN, platelets <0.5 x LLN, eosinophils >1.2 x ULN, activated partial thromboplastin time >1.1 x ULN, prothrombin time >1.1 x ULN, prothrombin intl. normalized ratio >1.1 x ULN; bilirubin/direct bilirubin/indirect bilirubin >1.5 x ULN, aspartate aminotransferase/alanine aminotransferase/gamma glutamyl transferase >3.0 x ULN, albumin <0.8 x LLN, urate >1.2 x ULN, bicarbonate >1.1 x ULN, triacylglycerol lipase >1.5 x ULN; urine hemoglobin/urine urobilinogen/urine nitrite/urine leukocyte esterase ≥1.
Time Frame: Baseline to Day 3
Population: All participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 3 | 4 | 5 | 6

7. Secondary Outcome: Number of Participants With Categorical Vital Signs Data
Description: Vital signs categorical criteria: 1) supine systolic blood pressure (SBP) <90 millimeters of mercury (mmHg); 2) supine diastolic blood pressure (DBP) <50 mmHg; 3) supine pulse rate <40 or >120 beats per minute (bpm); 4) change from baseline (increase or decrease) in supine SBP greater than or equal to (≥) 30 mmHg; 5) change from baseline (increase or decrease) in supine DBP ≥ 20 mmHg.
Time Frame: Baseline to Day 3
Population: All participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Pulse rate value <40 bpm | 0 | 0 | 0 | 0
  Pulse rate value >120 bpm | 0 | 0 | 0 | 0
  Sitting DBP value <50 mm Hg | 0 | 0 | 0 | 1
  Sitting DBP Change ≥ 20 mm Hg increase | 0 | 0 | 2 | 1
  Sitting DBP Change ≥ 20 mm Hg decrease | 0 | 0 | 0 | 0
  Sitting SBP value <90 mm Hg | 0 | 0 | 0 | 1
  Sitting SBP Change ≥ 30 mm Hg increase | 1 | 0 | 0 | 0
  Sitting SBP Change ≥ 30 mm Hg decrease | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Categorical Electrocardiogram (ECG) Data
Description: ECG categorical criteria: 1. PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization): a) greater than or equal to (≥) 300 millisecond (msec), b) ≥25% increase when baseline is > 200 msec or ≥50% increase when baseline is less than or equal to (≤) 200 msec.
  2. QRS interval (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization): a) ≥140 msec, b) ≥50% increase from baseline.
  3. QTcF interval (QT corrected using the Fridericia formula): a) >450 msec and ≤480 msec, b) >480 msec and ≤500 msec, c) >500 msec, d) >30 msec and ≤60 msec increase from baseline, e) >60 msec increase from baseline
Time Frame: Baseline to Day 3
Population: All participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  PR interval ≥300 msec | 0 | 0 | 0 | 0
  %Change in PR interval ≥25/50% | 0 | 0 | 0 | 1
  QRS interval ≥140 msec | 0 | 0 | 0 | 0
  %Change in QRS interval ≥50% | 0 | 0 | 0 | 0
  QTcF interval >450 and ≤480 msec | 0 | 1 | 1 | 3
  QTcF interval >480 and ≤500 msec | 0 | 0 | 0 | 0
  QTcF interval >500 msec | 0 | 0 | 0 | 0
  Change in QTcF interval >30 and ≤60 msec | 0 | 0 | 0 | 0
  Change in QTcF interval >60 msec | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Day 30
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 2/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Without Hepatic Impairment (N=6) | Mild Hepatic Impairment (N=6) | Moderate Hepatic Impairment (N=6) | Severe Hepatic Impairment (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT04604496/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT04604496/SAP_001.pdf